CLINICAL TRIAL: NCT00047983
Title: A Randomized Trial of Immunomodulating Diets With Arginine and Omega-3 Fatty Acids in Renal Transplant Recipients
Brief Title: Omega-3 Fatty Acids That Affect the Immune System in Kidney Transplant Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ID01
Record Dates: First submitted 2002-10-23; First posted 2002-10-24 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Kidney Diseases
Keywords: Kidney Transplantation; Fatty Acids, Omega-3; Erythrocyte Membrane; Graft Survival
MeSH Terms: conditions — Kidney Diseases | interventions — Rapeseed Oil; Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Controls and will receive no dietary supplements
- Arginine and Canola Oil (Experimental): Daily nutritional supplements of arginine and canola oil
  Interventions: Dietary Supplement: Canola oil; Dietary Supplement: Arginine
- Arginine and Coromega (Experimental): Daily nutritional supplements of arginine and Coromega
  Interventions: Dietary Supplement: Arginine; Dietary Supplement: Fish oil emulsion

INTERVENTIONS:
Dietary Supplement: Canola oil
  Arms: Arginine and Canola Oil
Dietary Supplement: Arginine
  Arms: Arginine and Canola Oil; Arginine and Coromega
Dietary Supplement: Fish oil emulsion
  Other Names: Coromega
  Arms: Arginine and Coromega

SUMMARY:
The purpose of this study is to evaluate the effectiveness of nutritional supplements in increasing the amount of omega-3 fatty acids (and arginine) in the red blood cell membranes and plasma of kidney transplant patients, and, secondarily, to compare patient compliance. The long-term goal of this study is to develop low risk therapies that will allow improved and lasting survival of donor tissue with minimal suppression of the immune system.

DETAILED DESCRIPTION:
Short-term survival rates of donor tissue after kidney transplantation have improved significantly in recent years because of improved immunosuppression. Rates of long-term tissue loss have changed less because of a high incidence of chronic rejection, infectious complications, and cardiovascular disease. Data suggest that both early and late complications might be reduced in transplant recipients by dietary intervention to raise levels of omega-3 fatty acids and arginine.

Prior to transplantation, participants are randomized to one of three groups. Group 1 participants serve as controls and receive no dietary supplements. Participants in Group 2 receive daily nutritional supplements of arginine and canola oil according to body weight. Group 3 participants receive daily nutritional supplements of arginine and a fish oil emulsion according to body weight. All participants receive a standard, low-fat dietary consultation. The status of participants is evaluated peri-transplant and at 1, 3, 6, and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease.
* Candidate to receive a living-related donor, living unrelated donor, or first cadaver kidney with at least 1 HLA mismatch.
* Negative crossmatch with the intended donor.
* Adults must have moderate to severe hypertension and/or take at least 1 medication for hypertension daily.
* Willingness to comply with the dietary supplements, including canola oil, a flavored drink mix, or an orange flavored pudding.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Women of childbearing age who are not willing or able to practice acceptable methods of contraception.
* HIV-positive.
* Positive test for HBV E-AG/DNA and HCV.
* Received an organ transplant or plan to receive a multiple organ transplant.
* Phenylketonuria.
* Participation in other investigational studies within 30 days of the renal transplant.
* Allergy or anaphylactic reactions to eggs or L-arginine.
* ABO blood incompatibility.
* Children who have previously received more than 5 blood transfusions.
* History of stroke.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Increases in omega-3 fatty acid levels in plasma and red blood cell membranes observed in each of the three omega-3 supplements used in this study

SECONDARY OUTCOMES:
Compliance rates observed in each of the three study groups

CONTACTS AND LOCATIONS:
Overall Officials: J. W. Alexander, MD, Principal Investigator — University of Cincinnati
Locations (4):
- United States (4):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] van der Heide JJ, Bilo HJ, Donker JM, Wilmink JM, Tegzess AM. Effect of dietary fish oil on renal function and rejection in cyclosporine-treated recipients of renal transplants. N Engl J Med. 1993 Sep 9;329(11):769-73. doi: 10.1056/NEJM199309093291105. PMID 8350886
- [Background] Daly JM, Lieberman MD, Goldfine J, Shou J, Weintraub F, Rosato EF, Lavin P. Enteral nutrition with supplemental arginine, RNA, and omega-3 fatty acids in patients after operation: immunologic, metabolic, and clinical outcome. Surgery. 1992 Jul;112(1):56-67. PMID 1377838
- [Background] Bower RH, Cerra FB, Bershadsky B, Licari JJ, Hoyt DB, Jensen GL, Van Buren CT, Rothkopf MM, Daly JM, Adelsberg BR. Early enteral administration of a formula (Impact) supplemented with arginine, nucleotides, and fish oil in intensive care unit patients: results of a multicenter, prospective, randomized, clinical trial. Crit Care Med. 1995 Mar;23(3):436-49. doi: 10.1097/00003246-199503000-00006. PMID 7874893
- [Background] Alexander JW, Levy A, Custer D, Valente JF, Babcock G, Ogle CK, Schroeder TJ. Arginine, fish oil, and donor-specific transfusions independently improve cardiac allograft survival in rats given subtherapeutic doses of cyclosporin. JPEN J Parenter Enteral Nutr. 1998 May-Jun;22(3):152-5. doi: 10.1177/0148607198022003152. PMID 9586793
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY352 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY352 — ImmPort study identifier is SDY352.
- Available data/document: Study Protocol: SDY352 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY352 — ImmPort study identifier is SDY352.
- Available data/document: Study summary, -design, -demographics, -lab tests, -study files: SDY352 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY352 — ImmPort study identifier is SDY352.